CLINICAL TRIAL: NCT04087915
Title: A Perspective, Cohort Study Assessing the Impact of Additional LDL-Cholesterol Reduction on Major Cardiovascular Events When Evolocumab is Used in Combination With Statin Therapy In Patients With High Risk Cardiovascular Disease
Brief Title: Further Cardiovascular Outcomes Research With PCSK9 Inhibition in Subjects With High Risk Coronary Artery Disease (FORWARD)
Acronym: FORWARD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Yujie Zhou, PhD,MD, Beijing Anzhen Hospital
Other Study IDs: FORWARD
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Dyslipidemia; High Risk Coronary Artery Disease
Keywords: High cholesterol; Treatment for high cholesterol; Lowering cholesterol; Lowering high cholesterol; Hypercholesterolemia
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia | interventions — evolocumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High risk coronary artery disease: Participants with high risk coronary artery disease.
  Interventions: Drug: Evolocumab

INTERVENTIONS:
Drug: Evolocumab — Participants received evolocumab 140 mg Q2W or 420 mg QM subcutaneous injections according to their own preference

SUMMARY:
The primary objective was to evaluate the effect of treatment with evolocumab on the risk for cardiovascular death, myocardial infarction, stroke, hospitalization for unstable angina, or coronary revascularization, whichever occurs first, in patients with high risk coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* Coronary artery disease at high risk (Syntax Score ≥ 33)
* Patients had to have a fasting LDL cholesterol level of 1.4 mmol per liter while they had been taken an optimized regimen of lipid-lowering therapy for at least 4 weeks, which was defined as preferably a high intensity statin but must have been at least atorvastatin at a dose of 20 mg daily or its equivalent, with or without ezetimibe.

Exclusion Criteria:

* New York Heart Association (NYHA) class III or IV, or last known left ventricular ejection fraction < 30%
* Uncontrolled hypertension
* Uncontrolled or recurrent ventricular tachycardia
* Untreated hyperthyroidism or hypothyroidism
* Homozygous familial hypercholesterolemia
* LDL or plasma apheresis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with high risk coronary artery disease
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-09-11 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of main adverse cardiovascular and cerebrovascular events (MACCE) | 1 year
  MACCE will include all-cause death, cardiovascular death, myocardial infarction, hospitalization for unstable angina, stroke, or coronary revascularization

SECONDARY OUTCOMES:
Reduction in LDL-C | up to 12 months
  Reduction in LDL-C reduction in LDL-C after 1 month, 3 months, 6 months and 12 months of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Yujie Zhou, PhD,MD, Study Chair — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided